CLINICAL TRIAL: NCT01545635
Title: RETIC Trial: Reversal of Trauma Induced Coagulopathy Using Coagulation Factor Concentrates or Fresh Frozen Plasma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Interim analysis (100 patients) revealed a possible harm to patients randomised to the fresh frozen plasma (FFP) treatment arm.
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Univ.-Doz. Dr. Petra Innerhofer, Principal Investigator, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RETIC
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Major Trauma
Keywords: Major trauma; Injury Severity Score; ISS > 15; clinical signs; risk of blood loss; coagulopathy; rotational thrombelastometry; ROTEM
MeSH Terms: conditions — Signs and Symptoms; Hemostatic Disorders | interventions — Fibrinogen; Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coagulation factor concentrates (Active Comparator)
  Interventions: Drug: Fibrinogen concentrate, Prothrombin complex concentrate and FXIII concentrate
- Fresh Frozen Plasma (Active Comparator)
  Interventions: Drug: Fresh Frozen Plasma blood type 0, A, B and AB

INTERVENTIONS:
Drug: Fibrinogen concentrate, Prothrombin complex concentrate and FXIII concentrate — Fibrinogen concentrate Dose: 50 mg/kg BW fibrinogen concentrate if FIBTEM A10<7mm Kind of application: Intravenously Frequency and rate of administration: Single-dose or repeated, each single vial (1g) over 5 min
  Prothrombin complex concentrate Dose: 20IE/kg BW PCC if EXTEM CT >90sec and FIBTEM A10>7mm Kind of application: Intravenously Frequency and rate of administration: Single-dose or repeated, each single dose over 10 min
  FXIII concentrate Dose: 20 IU/kg BW Fibrogammin® P will be administered with the second dose of fibrinogen concentrate (=100 mg/kg) and if FXIII decreases below 60% as detected by laboratory measurements.
  Kind of application: Intravenously Frequency and rate of administration: Single-dose or repeated, each single dose over 10 min
  Arms: Coagulation factor concentrates
Drug: Fresh Frozen Plasma blood type 0, A, B and AB — Fresh Frozen Plasma Dose: 15ml/kg BW if FibTEM A10 <7mm and/or ExTEM CT>90sec. Kind of application: Intravenously Frequency and rate of administration: Single-dose or repeated, each single U (200mL) over 5 min
  Arms: Fresh Frozen Plasma

SUMMARY:
Severe traumatized patients (ISS > 15) admitted to emergency department (ED) University Hospital Innsbruck with obvious bleeding and/or who are at risk for significant hemorrhage will be screened by rotational thrombelastometry (ROTEM) assays during ED treatment and subsequent surgical/radiological interventions for having coagulopathy (T0). If a patient meets the inclusion criteria (T1) and is recruited for the study, a first study related blood sample (40mL) will be drawn, and data collected. Subsequently, 100 patients will be randomized to receive Fibrinogen concentrate and/or Prothrombin complex concentrate and/or FXIII concentrate for reversal of coagulopathy, while the other 100 patients will receive fresh frozen plasma (FFP),respectively.

Treatment failure will be registered if bleeding persists and ROTEM parameters do not improve after two times dosages of study drug. In these cases haemostatic rescue therapy will be administered. CFC (fibrinogen concentrate and/or PCC, and/or FXIII concentrate) will be administered to patients randomized to receive FFP and FFP will be administered to patients of the CFC group.

In cases unresponsive to comprehensive treatment or normal ROTEM combined with diffuse bleeding, other haemostatic medications can be administered (e.g rFVIIa, DDAVP, VWF/FVIII concentrate) as judged by the anesthetist in charge. The need and type of any rescue therapy will be documented and a ROTEM will be performed thereafter.

At admission to ICU (T0 ICU), 24h (T24 ICU) and 48h(T48 ICU) thereafter further study related blood samples are drawn (40mL each).

The indications for transfusion of red blood cells or platelets, administration of antifibrinolytics, treatment of acidosis, hypothermia, hypocalcemia and volume replacement are similar for both groups and treatment is performed according to clinical routine.

Besides coagulation management during ED treatment until 24h on ICU, patient's care is not influenced by the study and follows clinical routine.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects =/> 18 years and =/< 80 years
2. Major trauma (ISS > 15)
3. Clinical signs of ongoing bleeding or patients who are at risk for significant haemorrhage assessed and judged by the ED team in charge of patient
4. Presence of coagulopathy defined by ROTEM assays as follows,

   * Patients with concomitant decreased fibrinogen polymerisation (ROTEM® FibTEM A10 of < 7 mm after 10 min)
   * Patients with concomitant decreased coagulation factor levels (ROTEM® ExTEM CT of > 90 sec)

Exclusion Criteria:

1. Lethal injury
2. CPR on the scene,
3. Isolated brain injury, burn injury
4. Avalanche injury
5. Administration of FFP or coagulation factor concentrates before ED admission
6. Delayed (> 6hours after trauma) admittance to ED
7. Known use of oral anticoagulants, or platelet aggregation inhibitors within 5 days before injury
8. Known history of severe allergic reaction to plasma products
9. Known history of congenital hemostasis disturbance, IgA or Protein C deficiency
10. Patients with a history of thromboembolic events or heparin induced thrombocytopenia (HIT) type 2 within the last year
11. Patients with a body weight < 45kg and > 150kg
12. Patients that are known to be pregnant
13. Jehova's Witness
14. Known participation in another clinical trial
15. Patient with known refusal of a participation in this clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Multiple Organ Failure (MOF) | Variable until 24h on ICU at the end of the IMP-administration
  Difference in the MOF as assessed by the Sequential Organ Failure Assessment score (SOFA) between treatment groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck / Department for Anesthesia and Intensive Care Medicine, Innsbruck, Tyrol, Austria

REFERENCES:
- [Derived] Innerhofer P, Fries D, Mittermayr M, Innerhofer N, von Langen D, Hell T, Gruber G, Schmid S, Friesenecker B, Lorenz IH, Strohle M, Rastner V, Trubsbach S, Raab H, Treml B, Wally D, Treichl B, Mayr A, Kranewitter C, Oswald E. Reversal of trauma-induced coagulopathy using first-line coagulation factor concentrates or fresh frozen plasma (RETIC): a single-centre, parallel-group, open-label, randomised trial. Lancet Haematol. 2017 Jun;4(6):e258-e271. doi: 10.1016/S2352-3026(17)30077-7. Epub 2017 Apr 28. PMID 28457980